CLINICAL TRIAL: NCT05253430
Title: Prognostic Implications of D1 vs D2 Lymphadenectomy in Gastric Cancer: a Propensity Score Matched Analysis
Brief Title: D1 vs D2 Lymphadenectomy in Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/115
Record Dates: First submitted 2022-01-13; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-12

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; lymphadenectomy; outcomes
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D1 lymph node dissection (LND): Patients with gastric cancer that underwent curative surgery with gastrectomy and D1 lymph node dissection
- D2 lymph node dissection (LND): Patients with gastric cancer that underwent curative surgery with gastrectomy and D2 lymph node dissection
  Interventions: Procedure: Lymphadenectomy type

INTERVENTIONS:
Procedure: Lymphadenectomy type — D1 vs D2 lymph node dissection
  Groups: D2 lymph node dissection (LND)

SUMMARY:
This study is a retrospective study with a propensity score-matched analysis in order to balance differences between patients with D1 and D2 lymphadenectomy for gastric cancer.The main aim is to analyse differences in the postoperative and oncological outcomes of patients with gastric cancer (GC) who underwent D1 and D2 gastrectomy.

DETAILED DESCRIPTION:
In this propensity score-matched analysis of 128 patients, D2 lymphadenectomy improved long-term outcomes compared with D1 in patients with curative intent surgery for gastric cancer except for the group of patients older than 75 years and with early tumors.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with GC stage I-III who underwent a curative gastrectomy +/- perioperative chemotherapy

Exclusion Criteria:

* patients with adenocarcinoma Siewert type I/II, palliative surgery, R1/R2 resections and pathological stage (pStage) IV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective study was carried out in all consecutive patients diagnosed with GC who underwent curative-intent surgery between April 1999 and October 2019
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 1990-04 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | percentage of patients without disease recurrence alive at 3 and 5 years after surgery
  Disease-free survival (DFS) was defined as the time from gastric surgery to the date of recurrence (locoregional, peritoneal recurrence and/or distant metastases).

SECONDARY OUTCOMES:
Overall survival | percentage of patients alive at 3 and 5 years after surgery
  Overall survival (OS) was defined as the time from the date of surgery to the date of death from any cause
Postoperative morbidity | from the surgery up to 90 days after the surgery
  Surgical complications were defined as any deviation from the normal postoperative course within 90 days after surgery, both during the hospital stay or after discharge.
Postoperative mortality | from the surgery up to 90 days after the surgery
  Mortality through post-operative follow-up

IPD SHARING:
Plan to Share IPD: No